CLINICAL TRIAL: NCT07125274
Title: Biomarker-guided Diagnosis of Tuberculosis
Brief Title: Sputum-free Diagnostis of TB
Acronym: TB_Diagnostics
Status: Recruiting | Type: Observational
Sponsor: Research Center Borstel (Other)
Responsible Party: Principal Investigator, Thomas Theo Brehm, Dr. med., Research Center Borstel
Other Study IDs: TBDiagnostics2025-101457-BO-ff
Record Dates: First submitted 2025-04-29; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis
Keywords: TB; diagnostics; sputum; sputum-free; transcriptomic; pathfast; CRISPR; stool; PCR
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with suspected TB
  Interventions: Diagnostic Test: Biomarker-guided diagnostic tests
- Other pulmonary infections (control group)
  Interventions: Diagnostic Test: Biomarker-guided diagnostic tests

INTERVENTIONS:
Diagnostic Test: Biomarker-guided diagnostic tests — mRNA-Signature from blood; immunophenotyping from blood; MBLA from sputum, PATHFAST-LAM and EclLAM from sputum, stool, urine; CRISPR-Cas from blood; stool PCR; QuantiFERON(R)-TB Gold Plus.

SUMMARY:
The aim of this study is to identify new biomarkers that enable reliable, non-invasive diagnosis of tuberculosis (TB), including in patients who are unable to produce sputum. The study analyzes biomaterials (blood, urine, stool, sputum) collected from patients with suspected TB. Various diagnostic methods are applied to assess the feasibility of individual and combined biomarker tests.

Participating patients will provide biomaterial samples (blood, urine, stool, sputum) once. No additional examinations or invasive procedures will be performed. Routine diagnostic procedures remain unaffected.

This is a single-center, prospective observational study. Patients are enrolled as part of their clinical care at the University Medical Center Hamburg-Eppendorf.

ELIGIBILITY:
Inclusion Criteria:

* Suspected pulmonary or extrapulmonary tuberculosis, or confirmed pulmonary or extrapulmonary tuberculosis with less than 7 days of anti-tuberculosis treatment, OR other pulmonary infection (control group).
* Age ≥ 18 years
* Ability to provide informed consent
* Willingness to participate in the study

Exclusion Criteria:

* Lack of ability to provide informed consent
* Age < 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years of age, including women of childbearing potential with or without contraception. Only adult patients capable of giving informed consent will be included; obtaining consent from legal guardians is not planned.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of biomarker-guided diagnosis of TB - mRNA signatures | From enrollment to the end of the first week of treatment
  Assessment of the feasibility of tuberculosis (TB) diagnostics based on mRNA signatures.
Feasibility of biomarker-guided diagnosis of TB - cellular immunology | From enrollment to the end of the first week of treatment
  Assessment of the feasibility of tuberculosis (TB) diagnostics based on cellular immunology.
Feasibility of biomarker-guided diagnosis of TB - PATHFAST-LAM | From enrollment to the end of the first week of treatment
  Assessment of the feasibility of tuberculosis (TB) diagnostics based on PATHFAST-LAM.
Feasibility of biomarker-guided diagnosis of TB - EclLAM | From enrollment to the end of the first week of treatment
  Assessment of the feasibility of tuberculosis (TB) diagnostics based on EclLAM assays.
Feasibility of biomarker-guided diagnosis of TB - cell-free Mycobacterium tuberculosis DNA | From enrollment to the end of the first week of treatment
  Assessment of the feasibility of tuberculosis (TB) diagnostics based on cell-free Mycobacterium tuberculosis DNA.
Feasibility of biomarker-guided diagnosis of TB - MBLA | From enrollment to the end of the first week of treatment
  Assessment of the feasibility of tuberculosis (TB) diagnostics based on Mycobacterial Load Assay (MBLA).
Feasibility of biomarker-guided diagnosis of TB - stool PCR | From enrollment to the end of the first week of treatment
  Assessment of the feasibility of tuberculosis (TB) diagnostics based on stool PCR testing.
Feasibility of biomarker-guided diagnosis of TB - composit | From enrollment to the end of the first week of treatment
  Assessment of the feasibility of tuberculosis (TB) diagnostics based on a combination of mRNA signatures, cellular immunology, PATHFAST-LAM and EclLAM assays, cell-free Mycobacterium tuberculosis DNA analysis, MBLA, stool PCR testing, and QuantiFERON®-TB Gold Plus testing.

SECONDARY OUTCOMES:
Exploratory Analysis of Biomarker Profiles and Their Clinical Associations | From enrollment to the end of the first week of treatment.
  Degree of correlation between the different biomarkers.
Exploratory Analysis of Biomarker Profiles and Their Clinical Associations | From enrollment to the end of the first week of treatment.
  Qualitative and quantitative characterization of differences in biomarker profiles between pulmonary and extrapulmonary tuberculosis.
Exploratory Analysis of Biomarker Profiles and Their Clinical Associations | From enrollment to the end of the first week of treatment.
  Qualitative and quantitative characterization of sex-specific differences in biomarker expression patterns.
Exploratory Analysis of Biomarker Profiles and Their Clinical Associations | From enrollment to the end of the first week of treatment.
  Degree of correlation between biomarkers and disease severity, as well as their potential prognostic value.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Lange, Prof. Dr. Dr. h.c., Study Chair — Clinical Infectious Diseases, Research Center Borstel, Leibniz Lung Center; Marylyn Martina Addo, Prof. Dr., Study Chair — Institute for Infection Research and Vaccine Development, University Medical Center Hamburg-Eppendorf; Stefan Schmiedel, Dr. med., Study Chair — Division of Infectious Diseases, I. Department of Internal Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany
Locations (1):
- Division of Infectious Diseases, I. Department of Internal Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, ICF
Time Frame: Starting mid 2027